CLINICAL TRIAL: NCT01651884
Title: High Definition-transcranial Direct Current Stimulation (HD-tDCS) for Stroke Rehabilitation
Brief Title: Effects of tDCS Versus HD-tDCS for Stroke Rehabilitation
Acronym: tDCS- Aphasia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Soterix Medical (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00015784; 1R41NS076123-01 (NIH)
Record Dates: First submitted 2012-07-19; First posted 2012-07-27 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Aphasia
Keywords: Stroke; Anomia
MeSH Terms: conditions — Stroke; Anomia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High-Definition tDCS (Experimental)
  Interventions: Device: HD-tDCS (Soterix)
- Sponge tDCS (Experimental)
  Interventions: Device: Transcranial Direct Current Stimulation (Neuroconn)

INTERVENTIONS:
Device: HD-tDCS (Soterix) — Subjects will be given individualized dose (number of electrodes and electrode placement) through High-Definition electrodes to target fMRI determined targets
  Other Names: Soterix Medical High-Definition M x N stimulator; Soterix Medical HDTargets
  Arms: High-Definition tDCS
Device: Transcranial Direct Current Stimulation (Neuroconn)
  Other Names: Neuroconn
  Arms: Sponge tDCS

SUMMARY:
The purpose of this study is to assess the changes in language processing of patients with chronic aphasia after receiving non-invasive brain stimulation.Previous research using traditional transcranial direct current stimulation (tDCS) using 2 sponge electrodes has shown that persons with aphasia show more improvement after treatment when that treatment is accompanied by brain stimulation. Traditional tDCS has recently been modified to deliver current to more specific locations in the brain. This new delivery method is called high-definition tDCS (HD-tDCS). It is not known whether traditional tDCS (more diffuse current delivery) or HD-tDCS (more focal current delivery) will be the better approach for enhancing treatment outcomes. To answer this question, computerized speech-language treatment will be administered during the application of the different forms of brain stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. one-time ischemic stroke in the left hemisphere
2. greater than 6-months post-stroke onset
3. between 25 and 80 years of age
4. aphasia diagnosis (as determined by pre-treatment language-based testing)
5. right-handed (before the stroke)
6. native speaker of English
7. ability to provide informed written or verbal consent

Exclusion Criteria:

1. clinically reported history of dementia, alcohol abuse, psychiatric disorder, traumatic brain injury, or extensive visual acuity or visual-spatial problems
2. factors contraindicative of tDCS administration (sensitive scalp, previous brain surgery)
3. prior history of epileptic or unprovoked seizures occurring during the previous 12 months.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julius Fridriksson, PhD, Principal Investigator — University of South Carolina